CLINICAL TRIAL: NCT02238938
Title: Piecemeal Versus En Bloc Resection of Large Rectal Adenomas -A Prospective, Randomized Multicenter Study
Brief Title: Piecemeal Versus En Bloc Resection of Large Rectal Adenomas
Acronym: PERLA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment of study patients
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Clinical Director, Department of Interdisciplinary Endoscopy, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERLA; PV 4580 (Registry Identifier: Ethics committee)
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Adenoma With Mild Dysplasia; Colorectal Adenoma With Severe Dysplasia; Colorectal Adenomatous Polyp; Colorectal Low Grade Intraepithelial Neoplasia; Colorectal High Grade Intraepithelial Neoplasia
Keywords: piecemeal polypectomy; piecemeal endoscopic mucosal resection (EMR); endoscopic submucosal dissection (ESD); endoscopic en-bloc resection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- en-bloc resection (Experimental): En- bloc resection is done after marking by use of different customary endoscopic knifes including combining devices as hybrid knife to cut down the lesion. After submucosal injection of liquid (saline or equivalent) to elevate the tissue it will be dissected and removed by a snare of adequate size solitarily. Since the aim of this method is the total resection basally and laterally, only one session is intended.
  Interventions: Procedure: en-bloc resection
- piecemeal resection (Active Comparator): Piecemeal resection will be done by snare following marking and submucosal injection of saline or equivalent liquids. Small leftover adenoma tissue will be resected thoroughly by snare or forceps. High resolution endoscopes are mandatory.
  After three months, an APC therapy will follow any piecemeal resection, if necessary, another resection of leftover adenoma will be done. This second session can be done by sigmoidoscopy.
  Interventions: Procedure: piecemeal resection

INTERVENTIONS:
Procedure: en-bloc resection — En- bloc resection after marking by use of different customary endoscopic knifes including combining devices as hybrid knife to cut down the lesion. After submucosal injection of liquid (saline or equivalent) to elevate the tissue it will be dissected and removed by a snare of adequate size solitarily.
  Other Names: endoscopic submucosal dissection; ESD
  Arms: en-bloc resection
Procedure: piecemeal resection — Piecemeal resection is done by snare after marking and submucosal injection of saline or equivalent liquids. Small leftover adenoma tissue will be resected thoroughly by snare or forceps.
  After three months, an APC therapy will follow any piecemeal resection, if necessary, another resection of leftover adenoma will be done.
  Other Names: piecemeal polypectomy; piecemeal endoscopic mucosal resection; piecemeal EMR
  Arms: piecemeal resection

SUMMARY:
Currently, colonoscopy is the safest way to detect bowel tumors and polyps, since these can be biopsied and removed in one working process. If the size of adenomas is larger than 2 cm, resections are usually done in a hospital setting. For the resection of large adenomas, different approaches can be used. The so-called piecemeal resection is done with snares, to cut off parts of the adenoma piece by piece until the whole adenoma is resected. This technique is the standard therapy, but is not required for very large adenomas, which can often show cell alterations that indicate cancer. Therefore these adenomas should be resected in one piece. This is done by the so-called en-bloc resection. For this kind of therapy, different endoscopic knifes are use to cut off the adenoma as a whole. Both resection techniques are done usually by previous injection of saline or other liquids to elevate the lesion from its bottom tissue.

Although the piecemeal resection of large adenoma is the standard therapy, it shows recurrence rates of 10 to 25%, which afford repeated therapies and follow up controls. En-bloc resections, though, are expected to have less recurrence rates but are much more complex to perform. They have higher complication rates especially in the West, where it has bee introduced only a couple of years ago.

The data situation regarding safety and efficacy of both therapies is low. This study is the first one ever to compare piecemeal EMR and ESD in a randomized way. The study might have influence on the logistics of future adenoma processing and patient flow.

DETAILED DESCRIPTION:
In 20 to 35% of colonoscopies due to symptoms or for prevention polyps, so-called adenoma, are found. Currently, colonoscopy is the best way to detect bowel tumors and polyps, since these can be biopsied and removed in one working process. If the size of adenoma is larger than 2 cm, resections are usually done in a hospital setting. Foremost for flat adenoma, the resection by snares piece by piece, the so-called piecemeal polypectomy, or piecemeal endoscopic mucosal resection (EMR), is state of the art. Resection will usually follow a submucosal saline injection (saline assisted polypectomy). Recurrences occur in 10 up to 25 %, requiring a reapplication of endoscopic therapy and follow up examinations.

Depending on the size of adenoma, increasing amounts of cell alterations of an advanced stage such as high grade dysplasia / intraepithelial neoplasia (HGIN) up to early cancer are found. In these cases, for histo-pathological and oncological reasons, a resection in a solitary manner (en-bloc resection) is necessary to evaluate the completeness of resection properly. Also, former studies showed that recurrence rate could be decreased considerably by en-bloc resections, since the aim is to perform a complete resection basally and laterally. New endoscopic techniques of en-bloc resections have been introduced since a couple of years, using several endoscopic knifes to cut adenoma down after submucosal injection of liquid and consecutively dissect it from the tissue underneath. This technique is mostly called endoscopic submucosal dissection (ESD), and, with not too large adenoma, can be combined with snare resection, too. The complexity of this method though is much larger than that of snare resection. Therefore, the western success rate is considerably less than in Japan, where it was developed first, and where higher numbers of cases exist in the upper GI tract as well as in the lower GI tract. All in all, the complication rate of en-bloc resection is higher than that of snare resection. Those complications, mostly perforations, are endoscopically controllable in most cases, though.

In comparison with Japan, Korea or China, early malign lesions oft he upper GI tract in the West are rare. Therefore, this study will be conducted on (colo)rectal lesions, which appear much more often in the West.

All in all, for efficacy (resection in total, number of recurrences) and risk (perforations), there is an indistinct data situation between piecemeal resection (EMR) and en-bloc resection (ESD). Up to now, no randomised comparing data exist. The planned study is the first randomised study between ESD and piecemeal EMR at all, since there are no studies been done for the upper GI tract, either. For reasons of complexity, ESD will conceivably remain a method for specialized centers, while piecemeal polypectomies are done in numerous hospitals. Therefore, the outcomes of this study will have influence on future logistics in polypectomies and flow of patients with large colorectal adenoma.

Piecemeal resection will be done by snare following marking and submucosal injection of saline or equivalent liquids. Small leftover adenoma tissue will be resected thoroughly by snare or forceps. High resolution endoscopes are mandatory.

After three months, an Argon plasma coagulation (APC) therapy will follow any piecemeal resection, if necessary, another resection of leftover adenoma will be done. This second session can be done by sigmoidoscopy.

En- bloc resection is done after marking by use of different customary endoscopic knifes including combining devices as hybrid knife to cut down the lesion. After submucosal injection of liquid (saline or equivalent) to elevate the tissue it will be dissected and removed by a snare of adequate size solitarily. Since the aim of this method is the total resection basally and laterally, only one session is intended.

Follow-up care: sigmoidoscopy after 6 and 18 months, colonoscopy after 36 months each after the end of the primary therapy session(s). Diagnostics will be done endoscopically and histologically of at least 6 biopsies if the size of lesion was up to 3 cm, and of at least 10 biopsies for larger lesions.

ELIGIBILITY:
Inclusion Criteria:

* patients with large non pedunculated colorectal adenomas designated for endoscopic resection up to 15 cm ab ano, length 2 cm to 5 cm, maximum hemicircumferential
* age > 18 years
* signed Informed Consent

Exclusion Criteria:

* adenomas smaller or larger than described above
* more than one large rectal adenoma
* adenomas with known or suspected carcinoma, proven by previous biopsies
* adenomas with known or suspected carcinoma that do not seem to be resectable by endoscopy, e.g. ulcers, suspected infiltration of submucosa after endoscopic or ultrasound diagnostics
* patients with chronic inflammatory bowel diseases
* severe general disease, including metastasising carcinomas
* coagulation abnormalities or anticoagulant drug use which make resection therapy impossible
* bad general state of health (American Society of Anesthesiologists Classification (ASA) IV or more)
* pregnancy and lactation
* recurrence or leftover dysplasia after extended endoscopic or surgical therapy (transanal endoscopic microsurgery (TEM))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
success rate of complete resection | 6 and 18 months after primary therapy
  success rate is confirmed by endoscopical diagnostics as well as histological diagnostics (at lest 6 biopsies in lesions up to 3 cm size, at least 10 biopsies in larger lesions). Patients with no complete resection will be treated further according to clinical requirement, depending on histology.

SECONDARY OUTCOMES:
en-bloc group: rate of R0 resections | timeline 0, day of en-bloc resection
  This parameter is regarding histopathology. Since piecemeal resections do not allow such a diagnosis, this parameter is only for the en-bloc resected group.
recurrence rate after complete adenoma resection | 36 months after initial resection
  Since early recurrences can evolve from leftover tumor cells and will become manifest after a time, the third control after two controls with negative biopsies.has been chosen to be the gold standard.
progress of therapy in patients with incomplete resection and recurrences | 36 months after initial resection
  patients will be treated further according to treatment standard depending on endoscopical and histological findings
differences in the subgroups of adenomas | 5 years
  size, shape according to nice classification, low-grade and high grade intraepithelial adenomas, sm1 carcinomas
required time for the initial procedure | timeline 0, day of initial resection
  for piecemeal resections including second procedure with APC therapy
complications including success of complication management | 5 years
  rate of complications that need intervention, e.g.
  * perforation (intra - and post procedural, surgery, additional procedures such as antibiotics, monitoring, intensive care
  * secondary haemorrhage (second look endoscopy, surgery)
  * infection
complications through patient sedation | timeline 0, day of initial resection
  depending on sedation standards of the participating centers
resolution of tumor board for post resections and outcomes of patients with carcinoma histology | 5 years
  patients with carcinoma histology will be discussed by a of tumor board

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Study Chair — University Hospital Eppendorf, Hamburg
Locations (6):
- Germany (5):
  - Sana Klinikum Lichtenberg, Berlin
  - Vivantes Wenckebach-Klinikum, Berlin
  - University Hospital Eppendorf, Hamburg
  - St. Bernward Krankenhaus, Hildesheim
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Risio M. The natural history of colorectal adenomas and early cancer. Pathologe. 2012 Nov;33 Suppl 2:206-10. doi: 10.1007/s00292-012-1640-6. PMID 22945585
- [Background] Lieberman DA, Weiss DG, Harford WV, Ahnen DJ, Provenzale D, Sontag SJ, Schnell TG, Chejfec G, Campbell DR, Kidao J, Bond JH, Nelson DB, Triadafilopoulos G, Ramirez FC, Collins JF, Johnston TK, McQuaid KR, Garewal H, Sampliner RE, Esquivel R, Robertson D. Five-year colon surveillance after screening colonoscopy. Gastroenterology. 2007 Oct;133(4):1077-85. doi: 10.1053/j.gastro.2007.07.006. PMID 17698067
- [Background] Saini SD, Kim HM, Schoenfeld P. Incidence of advanced adenomas at surveillance colonoscopy in patients with a personal history of colon adenomas: a meta-analysis and systematic review. Gastrointest Endosc. 2006 Oct;64(4):614-26. doi: 10.1016/j.gie.2006.06.057. PMID 16996358
- [Background] Stegeman I, de Wijkerslooth TR, Stoop EM, van Leerdam ME, Dekker E, van Ballegooijen M, Kuipers EJ, Fockens P, Kraaijenhagen RA, Bossuyt PM. Colorectal cancer risk factors in the detection of advanced adenoma and colorectal cancer. Cancer Epidemiol. 2013 Jun;37(3):278-83. doi: 10.1016/j.canep.2013.02.004. Epub 2013 Mar 9. PMID 23491770
- [Background] van Heijningen EM, Lansdorp-Vogelaar I, Kuipers EJ, Dekker E, Lesterhuis W, Ter Borg F, Vecht J, De Jonge V, Spoelstra P, Engels L, Bolwerk CJ, Timmer R, Kleibeuker JH, Koornstra JJ, van Ballegooijen M, Steyerberg EW. Features of adenoma and colonoscopy associated with recurrent colorectal neoplasia based on a large community-based study. Gastroenterology. 2013 Jun;144(7):1410-8. doi: 10.1053/j.gastro.2013.03.002. Epub 2013 Mar 7. PMID 23499951
- [Background] Jang JH, Balik E, Kirchoff D, Tromp W, Kumar A, Grieco M, Feingold DL, Cekic V, Njoh L, Whelan RL. Oncologic colorectal resection, not advanced endoscopic polypectomy, is the best treatment for large dysplastic adenomas. J Gastrointest Surg. 2012 Jan;16(1):165-71; discussion 171-2. doi: 10.1007/s11605-011-1746-9. Epub 2011 Nov 5. PMID 22058042
- [Background] Repici A, Hassan C, De Paula Pessoa D, Pagano N, Arezzo A, Zullo A, Lorenzetti R, Marmo R. Efficacy and safety of endoscopic submucosal dissection for colorectal neoplasia: a systematic review. Endoscopy. 2012 Feb;44(2):137-50. doi: 10.1055/s-0031-1291448. Epub 2012 Jan 23. PMID 22271024
- [Background] Farhat S, Chaussade S, Ponchon T, Coumaros D, Charachon A, Barrioz T, Koch S, Houcke P, Cellier C, Heresbach D, Lepilliez V, Napoleon B, Bauret P, Coron E, Le Rhun M, Bichard P, Vaillant E, Calazel A, Bensoussan E, Bellon S, Mangialavori L, Robin F, Prat F; SFED ESD study group. Endoscopic submucosal dissection in a European setting. A multi-institutional report of a technique in development. Endoscopy. 2011 Aug;43(8):664-70. doi: 10.1055/s-0030-1256413. Epub 2011 May 27. PMID 21623560
- [Background] Probst A, Pommer B, Golger D, Anthuber M, Arnholdt H, Messmann H. Endoscopic submucosal dissection in gastric neoplasia - experience from a European center. Endoscopy. 2010 Dec;42(12):1037-44. doi: 10.1055/s-0030-1255668. Epub 2010 Oct 22. PMID 20972955
- [Background] Ribeiro-Mourao F, Pimentel-Nunes P, Dinis-Ribeiro M. Endoscopic submucosal dissection for gastric lesions: results of an European inquiry. Endoscopy. 2010 Oct;42(10):814-9. doi: 10.1055/s-0030-1255778. Epub 2010 Sep 30. PMID 20886399
- [Background] Neuhaus H, Terheggen G, Rutz EM, Vieth M, Schumacher B. Endoscopic submucosal dissection plus radiofrequency ablation of neoplastic Barrett's esophagus. Endoscopy. 2012 Dec;44(12):1105-13. doi: 10.1055/s-0032-1310155. Epub 2012 Sep 11. PMID 22968641
- [Background] Probst A, Golger D, Anthuber M, Markl B, Messmann H. Endoscopic submucosal dissection in large sessile lesions of the rectosigmoid: learning curve in a European center. Endoscopy. 2012 Jul;44(7):660-7. doi: 10.1055/s-0032-1309403. Epub 2012 Apr 23. PMID 22528673
- [Background] Adler A, Roll S, Marowski B, Drossel R, Rehs HU, Willich SN, Riese J, Wiedenmann B, Rosch T; Berlin Private-Practice Gastroenterology Working Group. Appropriateness of colonoscopy in the era of colorectal cancer screening: a prospective, multicenter study in a private-practice setting (Berlin Colonoscopy Project 1, BECOP 1). Dis Colon Rectum. 2007 Oct;50(10):1628-38. doi: 10.1007/s10350-007-9029-y. PMID 17694415
- [Background] Redaelli A, Cranor CW, Okano GJ, Reese PR. Screening, prevention and socioeconomic costs associated with the treatment of colorectal cancer. Pharmacoeconomics. 2003;21(17):1213-38. doi: 10.2165/00019053-200321170-00001. PMID 14986736
- [Background] Soerjomataram I, Lortet-Tieulent J, Parkin DM, Ferlay J, Mathers C, Forman D, Bray F. Global burden of cancer in 2008: a systematic analysis of disability-adjusted life-years in 12 world regions. Lancet. 2012 Nov 24;380(9856):1840-50. doi: 10.1016/S0140-6736(12)60919-2. Epub 2012 Oct 16. PMID 23079588
- [Background] van den Broek FJ, de Graaf EJ, Dijkgraaf MG, Reitsma JB, Haringsma J, Timmer R, Weusten BL, Gerhards MF, Consten EC, Schwartz MP, Boom MJ, Derksen EJ, Bijnen AB, Davids PH, Hoff C, van Dullemen HM, Heine GD, van der Linde K, Jansen JM, Mallant-Hent RC, Breumelhof R, Geldof H, Hardwick JC, Doornebosch PG, Depla AC, Ernst MF, van Munster IP, de Hingh IH, Schoon EJ, Bemelman WA, Fockens P, Dekker E. Transanal endoscopic microsurgery versus endoscopic mucosal resection for large rectal adenomas (TREND-study). BMC Surg. 2009 Mar 13;9:4. doi: 10.1186/1471-2482-9-4. PMID 19284647
- [Background] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Background] Kim HH, Kim JH, Park SJ, Park MI, Moon W. Risk factors for incomplete resection and complications in endoscopic mucosal resection for lateral spreading tumors. Dig Endosc. 2012 Jul;24(4):259-66. doi: 10.1111/j.1443-1661.2011.01232.x. Epub 2012 Feb 7. PMID 22725112
- [Background] Kobayashi N, Yoshitake N, Hirahara Y, Konishi J, Saito Y, Matsuda T, Ishikawa T, Sekiguchi R, Fujimori T. Matched case-control study comparing endoscopic submucosal dissection and endoscopic mucosal resection for colorectal tumors. J Gastroenterol Hepatol. 2012 Apr;27(4):728-33. doi: 10.1111/j.1440-1746.2011.06942.x. PMID 22004124
- [Background] Ahlawat SK, Gupta N, Benjamin SB, Al-Kawas FH. Large colorectal polyps: endoscopic management and rate of malignancy: does size matter? J Clin Gastroenterol. 2011 Apr;45(4):347-54. doi: 10.1097/MCG.0b013e3181f3a2e0. PMID 20871408
- [Background] Ah Soune P, Menard C, Salah E, Desjeux A, Grimaud JC, Barthet M. Large endoscopic mucosal resection for colorectal tumors exceeding 4 cm. World J Gastroenterol. 2010 Feb 7;16(5):588-95. doi: 10.3748/wjg.v16.i5.588. PMID 20128027
- [Background] Hurlstone DP, Sanders DS, Cross SS, George R, Shorthouse AJ, Brown S. A prospective analysis of extended endoscopic mucosal resection for large rectal villous adenomas: an alternative technique to transanal endoscopic microsurgery. Colorectal Dis. 2005 Jul;7(4):339-44. doi: 10.1111/j.1463-1318.2005.00813.x. PMID 15932555
- [Background] Pigot F, Bouchard D, Mortaji M, Castinel A, Juguet F, Chaume JC, Faivre J. Local excision of large rectal villous adenomas: long-term results. Dis Colon Rectum. 2003 Oct;46(10):1345-50. doi: 10.1007/s10350-004-6748-1. PMID 14530673
- [Background] Doniec JM, Lohnert MS, Schniewind B, Bokelmann F, Kremer B, Grimm H. Endoscopic removal of large colorectal polyps: prevention of unnecessary surgery? Dis Colon Rectum. 2003 Mar;46(3):340-8. doi: 10.1007/s10350-004-6553-x. PMID 12626909
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Rosch T, Sarbia M, Schumacher B, Deinert K, Frimberger E, Toermer T, Stolte M, Neuhaus H. Attempted endoscopic en bloc resection of mucosal and submucosal tumors using insulated-tip knives: a pilot series. Endoscopy. 2004 Sep;36(9):788-801. doi: 10.1055/s-2004-825838. PMID 15326574
- [Background] Neuhaus H, Costamagna G, Deviere J, Fockens P, Ponchon T, Rosch T; ARCADE Group. Endoscopic submucosal dissection (ESD) of early neoplastic gastric lesions using a new double-channel endoscope (the "R-scope"). Endoscopy. 2006 Oct;38(10):1016-23. doi: 10.1055/s-2006-944830. PMID 17058167
- [Background] Adler A, Wegscheider K, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Gerber K, Stange G, Roll S, Gauger U, Wiedenmann B, Altenhofen L, Rosch T. Factors determining the quality of screening colonoscopy: a prospective study on adenoma detection rates, from 12,134 examinations (Berlin colonoscopy project 3, BECOP-3). Gut. 2013 Feb;62(2):236-41. doi: 10.1136/gutjnl-2011-300167. Epub 2012 Mar 22. PMID 22442161
- [Background] Adler A, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Scheel M, Schroder A, Yenerim T, Wiedenmann B, Gauger U, Roll S, Rosch T. Latest generation, wide-angle, high-definition colonoscopes increase adenoma detection rate. Clin Gastroenterol Hepatol. 2012 Feb;10(2):155-9. doi: 10.1016/j.cgh.2011.10.026. Epub 2011 Nov 2. PMID 22056301
- [Background] Adler A, Aschenbeck J, Yenerim T, Mayr M, Aminalai A, Drossel R, Schroder A, Scheel M, Wiedenmann B, Rosch T. Narrow-band versus white-light high definition television endoscopic imaging for screening colonoscopy: a prospective randomized trial. Gastroenterology. 2009 Feb;136(2):410-6.e1; quiz 715. doi: 10.1053/j.gastro.2008.10.022. Epub 2008 Oct 15. PMID 19014944
- [Background] Adler A, Pohl H, Papanikolaou IS, Abou-Rebyeh H, Schachschal G, Veltzke-Schlieker W, Khalifa AC, Setka E, Koch M, Wiedenmann B, Rosch T. A prospective randomised study on narrow-band imaging versus conventional colonoscopy for adenoma detection: does narrow-band imaging induce a learning effect? Gut. 2008 Jan;57(1):59-64. doi: 10.1136/gut.2007.123539. Epub 2007 Aug 6. PMID 17681999
- [Background] Pohl H, Aschenbeck J, Drossel R, Schroder A, Mayr M, Koch M, Rothe K, Anders M, Voderholzer W, Hoffmann J, Schulz HJ, Liehr RM, Gottschalk U, Wiedenmann B, Rosch T. Endoscopy in Barrett's oesophagus: adherence to standards and neoplasia detection in the community practice versus hospital setting. J Intern Med. 2008 Oct;264(4):370-8. doi: 10.1111/j.1365-2796.2008.01977.x. Epub 2008 May 15. PMID 18482289
- [Background] Meining A, Ott R, Becker I, Hahn S, Muhlen J, Werner M, Hofler H, Classen M, Heldwein W, Rosch T. The Munich Barrett follow up study: suspicion of Barrett's oesophagus based on either endoscopy or histology only--what is the clinical significance? Gut. 2004 Oct;53(10):1402-7. doi: 10.1136/gut.2003.036822. PMID 15361485
- [Background] Heldwein W, Dollhopf M, Rosch T, Meining A, Schmidtsdorff G, Hasford J, Hermanek P, Burlefinger R, Birkner B, Schmitt W; Munich Gastroenterology Group. The Munich Polypectomy Study (MUPS): prospective analysis of complications and risk factors in 4000 colonic snare polypectomies. Endoscopy. 2005 Nov;37(11):1116-22. doi: 10.1055/s-2005-870512. PMID 16281142